CLINICAL TRIAL: NCT01757444
Title: Clinical Benefits and Tolerance to a New Ventilatory Mode in Patients With Obesity Hypoventilation Syndrome (OHS).
Brief Title: Non Invasive Ventilation : Efficacy of a New Ventilatory Mode in Patients With OHS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche (Other)
Responsible Party: Principal Investigator, DELRIEU Jacqueline, Coordinator, Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2012 - A00731 - 42; EVAL CLIN - VENTILATEUR (Other: ANTADIR)
Record Dates: First submitted 2012-12-17; First posted 2012-12-31 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Obesity Hypoventilation Syndrome
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BiPAP - A40 (Experimental): BiPAP with AVAPS AE mode
  Interventions: Device: BiPAP - A40
- BiPAP- ST (Active Comparator): Patients receiving BiPAP- ST at home
  Interventions: Device: BiPAP - ST

INTERVENTIONS:
Device: BiPAP - A40 — Patients receiving BiPAP AVAPS - AE ventilatory mode at home
  Arms: BiPAP - A40
Device: BiPAP - ST — Patients receiving BiPAP- ST mode at home.
  Arms: BiPAP- ST

SUMMARY:
In 2012, it has announced the availability of the new ventilator (BiPAP- A40), which could offer potential advantages over fixed level pressure support, in particular, in patients with obesity hypoventilation syndrome (OHS). One of the key benefits of the BiPAP A40 is an innovative ventilation mode called AVAPS-AE, which automatically maintains airway patency while delivering the correct level of ventilation each user requires, whatever their body position or sleep stage. AVAPS-AE mode is also aimed to help the clinicians during the initial titration of therapy, while providing long term comfort and assuring therapy compliance. However, studies on the physiologic and clinical effects have not yet been performed. The aim of our singled-blind randomised multicentre controlled trial is to prospectively investigate the effects of BiPAP with the spontaneous/timed (S/T) or the AVAPS-AE ventilation mode over 8 weeks on sleep quality, ventilation pattern, gas exchange, symptoms, body composition, level of physical activity and health-related quality of life in OHS patients.

DETAILED DESCRIPTION:
Efficacy on sleep quality, symptoms, physical activity and quality of life

ELIGIBILITY:
Inclusion Criteria:

* Man or woman, stable patient with obesity hypoventilation syndrome, naives of non invasive ventilation.
* PaCO2 ≥ 45 mmHg.
* PaO2 < 70 mmHg
* BMI ≥ 30Kg. m2

Exclusion Criteria:

* Chronic obstructive pulmonary disease
* Neuromuscular disease
* Scoliosis
* Cardiac insufficiency
* Significant psychiatric disease
* Sleep apnea syndrome with central apnea index > 10%
* Treatment with benzodiazepines at the inclusion

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-06; Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
CHANGE IN SLEEP QUALITY | Day 1 and Day 61
  Sleep stage, micro arousals, apnea/hypopnea index...

SECONDARY OUTCOMES:
CHANGE IN GAZ EXCHANGE | Day 1 and Day 61

OTHER OUTCOMES:
CHANGE IN QUALITY OF LIFE/ LEVEL OF PHYSICAL ACTIVITY/ BODY COMPOSITION | Day 1 and Day 61

CONTACTS AND LOCATIONS:
Overall Officials: Jean-François MUIR, Pr, Principal Investigator — Association Nationale pour les Traitements A Domicile, les Innovations et la Recherche
Locations (11):
- France (11):
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier de Béziers, Béziers
  - Hôpital Haut- Lévêque, Bordeaux
  - Centre Hospitalier de Cannes, Cannes
  - Clinique du Parc, Castelnau-le-Lez
  - Hôpital du Bocage, Dijon
  - Hôpital Michallon, Grenoble
  - Hôpital Pitié-Salpêtrière, Paris
  - Hôpital La Milétrie, Poitiers
  - Hôpital de Bois Guillaume, Rouen
  - Hôpital Larrey, Toulouse